CLINICAL TRIAL: NCT01855438
Title: Increasing Communication About Live Donor Kidney Transplant: A Proof of Concept
Brief Title: Increasing Communication About Live Donor Kidney Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HM12097; PD302305 (Other: VCU)
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Kidney Transplant Candidates
Keywords: Live donor kidney transplantation; Living donation; Patient education; Kidney transplant candidates

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): Kidney transplant candidates randomized to this arm will receive only the education provided by the transplant center. After data collection activities have concluded, transplant candidates in this arm will be offered the opportunity to attend a program session.
- Living Donor Transplant Education 1 (Experimental): Participants randomized to Living Donor Transplant Education 1 will receive education on living donor kidney transplantation and its discussion.
  Interventions: Behavioral: Living Donor Transplant Education
- Living Donor Transplant Education 2 (Experimental): Participants randomized to Living Donor Transplant Education 2 will receive education on living donor kidney transplantation and its discussion; they will also have the opportunity to practice discussing living kidney transplantation with simulated patients portraying participants' conversational partners.
  Interventions: Behavioral: Living Donor Transplant Education

INTERVENTIONS:
Behavioral: Living Donor Transplant Education — The Living Donor Transplant Education informs kidney transplant candidates about living donor transplants and provides guidance in broaching and maintaining discussion about the topic.
  Arms: Living Donor Transplant Education 1; Living Donor Transplant Education 2

SUMMARY:
This study will test the efficacy of a communication intervention intended to increase and improve kidney transplant candidates' communication about live donor kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Wait listed for kidney transplantation in active status (i.e., status 1 or 2)
* Adult (at least 18 years of age)
* English speaking
* Capable of making medical decisions (i.e., not cognitively impaired)
* Non-institutionalized

Exclusion Criteria:

* Not listed for kidney transplantation or wait listed, but not in active status
* Under 18 years of age
* Non-English speaking
* Cognitively impaired
* Institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2013-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in the number of individuals screened as potential living donors | Upon enrollment (baseline); 1 month post; 3 months post
  1 self-reported item

SECONDARY OUTCOMES:
Change in intentions to discuss live donor kidney transplantation | Upon enrollment (baseline); 1 month post; 3 months post
  3-item, 7-point Likert-type scale
Change in engagement in discussion about live donor kidney transplantation | Upon enrollment (baseline); 1 month post; 3 months post
  2 self-reported items: whether live donor kidney transplantation was discussed (yes/no) and number of discussions held
Change in the number of living donor kidney transplants performed | At study commencement; after all program sessions (interventions) are completed; at study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Traino, PhD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States